CLINICAL TRIAL: NCT04539314
Title: Dexmedetomidine as an Adjuvant to Bupivacaine in Unilateral Transversus Abdominis Plane Block in Pediatrics
Brief Title: Unilateral Transversus Abdominis Plane Block in Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, haidy salah mansour, Professor, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 274:7/2019
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Unilateral TAP Block in Pediatric Patients Undergoing Lower Abdominal Surgery
MeSH Terms: interventions — Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): TAP block will be performed using (0.5 ml/ kg bupivacaine 0.25%)
  Interventions: Drug: Bupivacain
- Dexmedetomidine 0.5 μg group (Active Comparator): TAP block will be performed using (0.5 ml/ kg bupivacaine 0.25%) plus dexmedetomidine 0.5 μg / kg as an adjuvant
  Interventions: Drug: Dexmedetomidine o.5 μg
- Dexmedetomidine 1 μg group (Active Comparator): TAP block will be performed using (0.5 ml/ kg bupivacaine 0.25%) plus dexmedetomidine 1 μg / kg as an adjuvant
  Interventions: Drug: Dexmedetomidine 1 μg

INTERVENTIONS:
Drug: Bupivacain — We will carry out the TAP block using 0.5 ml/ kg bupivacaine 0.25%
  Arms: Control group
Drug: Dexmedetomidine o.5 μg — We will carry out the TAP block using using 0.5 ml/ kg bupivacaine 0.25% with dexmedetomidine 0.5 μg / kg
  Arms: Dexmedetomidine 0.5 μg group
Drug: Dexmedetomidine 1 μg — We will carry out the TAP block using using 0.5 ml/ kg bupivacaine 0.25% with dexmedetomidine 1 μg / kg
  Arms: Dexmedetomidine 1 μg group

SUMMARY:
the present study was designed to compare the efficacy and safety of two different doses of dexmedetomidine as an adjuvant to bupivacaine in unilateral TAP block in pediatric patients undergoing lower abdominal surgery.

DETAILED DESCRIPTION:
After insertion of venous access, all children received premedication in the form of atropine at a dose of 0.01-0.02 mg/kg. Perioperative monitoring included continuous ECG, pulse oximetry and non-invasive arterial blood pressure. Baseline reading of heart rate, mean arterial blood pressure was recorded after monitor attachment.

General anesthesia will be induced using propofol 1.5-2.5 mg/kg over 20-30 s as tolerated, atracurium 0.5 mg/kg to facilitate endotracheal intubation. Anesthesia will be maintained using isoflurane (1 MAC) and atracurium 0.1 mg/kg supplements will be given to maintain muscle relaxation.

TAP block will be performed in All patients immediately after induction patients will be allocated randomly into three equal groups, 30 patients in each as the following.

Group 1 (control group) TAP block will be performed using (0.5 ml/ kg bupivacaine 0.25%) Group 2 We will carry out TAP block using the same dose of bupivacaine in the control group plus dexmedetomidine 0.5 μg / kg as an adjuvant Group (3) In this participants dexmedetomidine in dose 1 μg / kg will be given as an adjuvant to the control dose of bupivacaine in the TAP block TAP block procedure With the patient in the supine position, the site of the ultrasound and needle entry was sterilized. The TAP block will be performed laterally behind the midaxillary line between the iliac crest and the most inferior extent of the ribs. The plane between the internal oblique and transversus abdominis muscle located around the midaxillary line with the probe transverse to the abdomen. Anteriorly, the needle passes to come perpendicular to the ultrasound beam and placed between transversus and internal oblique posterior to the midaxillary line. Then, the local anesthetic will be injected. (Al-Sadek et al.,2014).

The procedure will be performed immediately after induction of anesthesia by candidate anesthesiologist who is not aware of group allocation.

After completion of surgical procedure anesthesia will be discontinued, muscle relaxant reversed using atropine 0.02 mg/kg and 0.05 mg/kg of neostigmine, extubated, and transferred to PACU.

Parameters will be assessed

• Quality of analgesia will be assessed immediately postoperatively and then at 2, 4, 8, 12 and 24 h postoperatively using FLACC scale (face,leg,activity,cry and consolability).

Time to the first analgesic requirement will be recorded from immediately postoperative to the time of FLACC score >6. Acetaminophen (perfalgan) 15 mg/kg IV will be given as rescue analgesia for patients if FLACC score >6 and total dose of acetaminophen will be recorded.

• Hemodynamic data including heart rate (HR) and mean arterial blood pressure (MAP).

Intraoperative any increase in heart rate and or mean arterial blood pressure by more than 20% of baseline values in response to surgical stimulus or thereafter throughout the whole operation warranted administration of intravenous fentanyl (0.5 μg/kg).

* postoperative complication including postoperative hypotension or bradycardia (decrease in MAP or HR by more than 20% of baseline value), postoperative nausea and vomiting (PONV)
* length of hospital stays, and patients or parents' satisfaction assessed on a 5-point scale (Al-Sadek et al.,2014) 1-completely dissatisfied, 2-dissatisfied, 3-not satisfied nor dissatisfied, 4- satisfied 5-completely satisfied

ELIGIBILITY:
Inclusion Criteria:

* ASA class I or II, aged from 1-7 years old undergoing any lower abdominal surgery that requires skin incision in one side of midline of the anterior abdominal wall

Exclusion Criteria:

* Participants refusing regional block and those having bleeding disorders, skin lesions or wounds at the site of proposed needle insertion, evidence of peritonitis, septicemia and hepatic disease or enlargement in addition to those who required emergency procedures or operations that requires exploratory longitudinal midline incision were excluded from the study

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-12-26 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Quality of analgesia | 24 hours after block
  Quality of analgesia will be assessed by using FLACC scale (face,leg,activity,cry and consolability)

SECONDARY OUTCOMES:
postoperative complication | For 24 hours after surgery
  postoperative complication including postoperative hypotension or bradycardia (decrease in MAP or HR by more than 20% of baseline value), postoperative nausea and vomiting (PONV)
parents' satisfaction | 24 hours
  parents' satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Amany khairy Abo el-hussein, Cairo, Minya Governorate, Egypt